CLINICAL TRIAL: NCT04827238
Title: Standardized Invasive Hemodynamics for Monitoring Acute and Long Term Valve Performance in Patients With Elevated Gradients Post Transcatheter Aortic Valve Replacement
Brief Title: Standardized Invasive Hemodynamics for Elevated Gradients Post TAVR (DISCORDANCE TAVR)
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Principal Investigator, David Wood, Clinical Professor, University of British Columbia
Other Study IDs: H21-00824
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Aortic Stenosis; Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with Elevated Gradients Post Transcatheter Aortic Valve Replacement: Patients who have an echocardiographic transaortic mean gradient ≥ 20mmHg OR VARC-3 criteria for ≥ moderate hemodynamic valve deterioration post TAVR on any TTE > 1 month post-TAVR
  Interventions: Diagnostic Test: Standardized Invasive Hemodynamics

INTERVENTIONS:
Diagnostic Test: Standardized Invasive Hemodynamics — The SIH technique is a standardized, reproducible and efficient way of obtaining hemodynamic measurements.

SUMMARY:
The DISCORDANCE TAVR study will determine the discordance between echocardiography-derived and invasive transaortic gradients, as determined by a consistent and reproducible technique (Standardized Invasive Hemodynamics) post-TAVR.

DETAILED DESCRIPTION:
Since the introduction of Doppler echocardiography, non-invasive estimation of aortic valve gradients through modification and simplification of the Bernoulli equation and derivation of the AVA, via the continuity equation, have become the primary method to assess the severity of AS.

The utility of echocardiography to successfully determine aortic valve gradients and AVA has been established in the presence of AS, and such observations have been extrapolated to prosthetic valves. However, several reports following SAVR and TAVR for both native and valve-in-valve have demonstrated significant discordance between echocardiography-derived and direct invasive measurements of aortic valve mean gradients.

The indexed AVA (iAVA) is derived from the stroke volume indexed to the BSA. The stroke volume index (SVI) divided by the Doppler velocity time integral of the continuous wave aortic valve spectral profile, is used to determine the presence of severe PPM. As such, a low iAVA may occur due to a low flow state defined by a reduced SVI (<35 ml/m2) or a reduced stroke flow rate (< 200 ml/second) and calculated by dividing the SV by the ejection time spuriously increasing the incidence of severe PPM. A low indexed effective orifice area due to a low SVI, in the absence of intrinsic PPM, has been referred to as "pseudo-severe PPM", but the impact of flow state on PPM has not been described.

Nonetheless, echocardiographic thresholds for the evaluation of prosthetic valve performance after TAVR have been widely adopted: mean-gradient > 20mmHg, severe PPM as defined by an iAVA < 0.65 cm2/m2, and AR, including paravalvular and transvalvular AR of moderate or greater severity. These criteria are suggested to indicate procedural success and predict long-term clinical outcomes (12). Practically many centers utilize an echocardiography-derived mean gradient for the follow-up of transcatheter heart valves. While the association of at least moderate paravalvular AR with mortality has been consistently demonstrated, there remains uncertainty regarding the clinical impact of severe PPM as determined by index echocardiography. Furthermore, the magnitude of discordance between echocardiography-derived and invasive aortic valve mean-gradients post TAVR is unknown and it remains unclear how to reconcile measurement discordances in clinical practice. These potential differences may have an important impact on patient management post TAVR.

The DISCORDANCE TAVR study will determine the discordance between echocardiography-derived and invasive transaortic gradients, as determined by a consistent and reproducible technique (Standardized Invasive Hemodynamics) post-TAVR.

ELIGIBILITY:
Inclusion Criteria:

* Echocardiographic transaortic mean gradient ≥ 20mmHg OR VARC-3 criteria for ≥ moderate hemodynamic valve deterioration post TAVR on any TTE > 1 month post-TAVR
* Consensus by the Heart Team that the patient is suitable for Standardized Invasive Hemodynamics (SIH).

Exclusion Criteria:

* CT demonstrating leaflet thrombosis or hypoattenuated leaflet thickening (HALT)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients > 1 month post-transcatheter aortic valve replacement
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Transaortic valve gradients | 30 days
  Transaortic valve gradients measured by echocardiography and direct invasive methods
Transaortic mean gradient reclassification | 30 days
  Proportion of patients reclassified to a transaortic mean gradient < 20mmHg using direct invasive methods
VARC-3 hemodynamic valve deterioration reclassification | 30 days
  Proportion of patients reclassified to ≤ moderate VARC-3 hemodynamic valve deterioration using direct invasive methods, including mean gradient and valve area, compared to echocardiography
Patient-Prosthesis Mismatch (PPM) reclassification | 30 days
  Proportion of patients with echocardiographic severe PPM reclassified as non-severe PPM using direct invasive methods

SECONDARY OUTCOMES:
Total procedure time | 30 days
  Total procedure time (mins) to complete standardized invasive hemodynamics
Risks of procedural complications | 30 days
  Evaluate risks of procedural complications associated with direct-invasive hemodynamics

CONTACTS AND LOCATIONS:
Overall Officials: David Wood, MD, Principal Investigator — University of British Columbia
Locations (9):
- United States (6):
  - PIMA Heart Centre, Tucson, Arizona
  - Tenet Health, Boca Raton, Florida
  - eCommunity, Indianapolis, Indiana
  - Community Hospital, Munster, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - William Beaumont Hospital, Southfield, Michigan
- Canada (3):
  - Vancouver General Hospital, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia
  - McMaster University, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No